CLINICAL TRIAL: NCT02920983
Title: A Clinical Comparison of Three Soft Daily Disposable Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: EX-MTKG-74 (C16-596)
Record Dates: First submitted 2016-09-29; First posted 2016-09-30 (Estimated); Results first posted 2019-06-26 (Actual); Last update posted 2019-10-17 (Actual); Status verified 2019-10

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- somofilcon A (Active Comparator): Subjects are randomized to wear somofilcon A for one week during the cross over study.
  Interventions: Device: somofilcon A
- nelfilcon A II 2 (Active Comparator): Subjects are randomized to wear nelfilcon A II 2 for one week during the cross over study.
  Interventions: Device: nelfilcon A II 2
- omafilcon A ll 2 (Active Comparator): Subjects are randomized to wear omafilcon A ll 2 for one week during the cross over study.
  Interventions: Device: omafilcon A ll 2

INTERVENTIONS:
Device: somofilcon A — contact lens
  Arms: somofilcon A
Device: nelfilcon A II 2 — contact lens
  Arms: nelfilcon A II 2
Device: omafilcon A ll 2 — contact lens
  Arms: omafilcon A ll 2

SUMMARY:
This study aims to compare the clinical performance of the somfilcon A, nelfilcon A II 2 and omafilcon A II 2 daily disposable contact lenses.

DETAILED DESCRIPTION:
This will be a randomised, subject-masked, crossover, bilateral study, controlled by cross comparison. Fifty subjects will use each lens type for a week in random sequence. Follow-up visits for each lens will be performed after one week of wear. Lenses will be worn on a daily wear, daily disposable wear schedule.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will only be eligible for the study if:

  1. They are of legal age (18) and capacity to volunteer.
  2. They understand their rights as a research subject and are willing and able to sign a Statement of Informed Consent.
  3. They are willing and able to follow the protocol.
  4. They agree not to participate in other clinical research for the duration of this study.
  5. They have a contact lens spherical prescription between -1.00 to - 6.00D (Diopters) (inclusive)
  6. They have a spectacle cylindrical correction of -0.75D or less in each eye.
  7. At dispensing, they can attain at least 0.10 logMAR distance high contrast visual acuity in each eye with the study lenses within the available power range.
  8. They currently use soft contact lenses or have done so in the previous six months.
  9. They are willing to comply with the wear schedule (at least five days per week and for at least eight hours per day).

Exclusion Criteria:

* Subjects will not be eligible to take part in the study if:

  1. They have an ocular disorder which would normally contra-indicate contact lens wear.
  2. They have a systemic disorder which would normally contra-indicate contact lens wear.
  3. They are using any topical medication such as eye drops or ointment.
  4. They have had cataract surgery.
  5. They have had corneal refractive surgery.
  6. They have any corneal distortion resulting from previous hard or rigid lens wear or have keratoconus.
  7. They are pregnant or breast-feeding.
  8. They have any ocular abnormality which would, in the opinion of the investigator, normally contraindicate contact lens wear.
  9. They have any infectious disease which would, in the opinion of the investigator, contraindicate contact lens wear or pose a risk to study personnel; or they have any immunosuppressive disease (e.g. HIV), or a history of anaphylaxis or severe allergic reaction.
  10. They have taken part in any other contact lens or care solution clinical trial or research, within two weeks prior to starting this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2016-09; Primary Completion 2016-11 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carole Maldonado-Codinal, PhD, FAAO, Principal Investigator — Eurolens Research, University of Manchester
Locations (1):
- Eurolens Research - The University of Manchester, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 55 subjects were recruited for the study, 51 subjects were enrolled and 50 subjects completed the initial follow up visit.
Pre-assignment Details: Subjects are randomized to wear each lens brand for one week in a random sequence.
Groups:
- Somofilcon A, Nelfilcon A II 2, Omafilcon A II 2: Subjects are randomized to wear somofilcon A pair of lenses for one week during the crossover study then nelfilcon A II2, then omafilcon A II 2 lenses for one week each.
- Somofilcon A, Omafilcon A II 2, Nelfilcon A II 2: Subjects are randomized to wear somofilcon A pair of lenses for one week during the cross-over study then omafilcon A II 2, then nelfilcon A II 2 lenses for one week each.
- Nelfilcon A II 2, Somofilcon A, Omafilcon A II 2: Subjects are randomized to wear nelfilcon A II 2 pair of lenses for one week during the cross-over study then Somofilcon A, then Omafilcon A II 2 lenses for one week each.
- Nelfilcon A II 2, Omafilcon A II 2, Somofilcon A: Subjects are randomized to wear nelfilcon A II 2 pair of lenses for one week during the cross-over study then Omafilcon A II 2, then Somofilcon A, lenses for one week each.
- Omafilcon A II 2, Nelficon A II 2, Somofilcon A: Subjects are randomized to wear omafilcon A II 2 pair of lenses for one week during the cross-over study then nelfilcon A II 2, then Somofilcon A lenses for one week each.
- Omafilcon A II 2, Somofilcon A, Nelfilcon A II 2: Subjects are randomized to wear omafilcon A II 2 pair of lenses for one week during the cross-over study then Somofilcon A, then nelfilcon A II 2 lenses for one week each.
Period: Dispense 1
Arm/Group | Somofilcon A, Nelfilcon A II 2, Omafilcon A II 2 | Somofilcon A, Omafilcon A II 2, Nelfilcon A II 2 | Nelfilcon A II 2, Somofilcon A, Omafilcon A II 2 | Nelfilcon A II 2, Omafilcon A II 2, Somofilcon A | Omafilcon A II 2, Nelficon A II 2, Somofilcon A | Omafilcon A II 2, Somofilcon A, Nelfilcon A II 2
Started | 8 | 10 | 7 | 6 | 13 | 7
Completed | 8 | 10 | 7 | 6 | 12 | 7
Not Completed | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Unacceptable Lens Fit | 0 | 0 | 0 | 0 | 1 | 0
Period: Dispense 2
Arm/Group | Somofilcon A, Nelfilcon A II 2, Omafilcon A II 2 | Somofilcon A, Omafilcon A II 2, Nelfilcon A II 2 | Nelfilcon A II 2, Somofilcon A, Omafilcon A II 2 | Nelfilcon A II 2, Omafilcon A II 2, Somofilcon A | Omafilcon A II 2, Nelficon A II 2, Somofilcon A | Omafilcon A II 2, Somofilcon A, Nelfilcon A II 2
Started | 8 | 10 | 7 | 6 | 13 | 7
Completed | 7 | 10 | 7 | 6 | 12 | 7
Not Completed | 1 | 0 | 0 | 0 | 1 | 0
Not completed — Unscceptable lens fit | 1 | 0 | 0 | 0 | 1 | 0
Period: Dispense 3
Arm/Group | Somofilcon A, Nelfilcon A II 2, Omafilcon A II 2 | Somofilcon A, Omafilcon A II 2, Nelfilcon A II 2 | Nelfilcon A II 2, Somofilcon A, Omafilcon A II 2 | Nelfilcon A II 2, Omafilcon A II 2, Somofilcon A | Omafilcon A II 2, Nelficon A II 2, Somofilcon A | Omafilcon A II 2, Somofilcon A, Nelfilcon A II 2
Started | 8 | 10 | 7 | 6 | 13 | 7
Completed | 7 | 9 | 7 | 6 | 12 | 7
Not Completed | 1 | 1 | 0 | 0 | 1 | 0
Not completed — Unacceptable Lens Fit | 1 | 1 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: 55 subjects were recruited for the study with 50 subjects completing initial follow up visit. 5 subjects were ineligible to be dispensed with lenses for sphere out of range or cylinder out of range.
Groups:
- Overall Study: Total participants
Arm/Group | Overall Study
Number analyzed (Participants) | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.6 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 20

OUTCOME MEASURES:

1. Primary Outcome: Ocular Physiology
Description: Ocular physiology assessment of by biomicroscopy (Scale 0-4, 0.25 steps, 0=normal, 4=severe).
Time Frame: 1 week
Population: Protocol deviations and discontinuations account for difference in analysis population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Somofilcon A | Nelfilcon A II 2 | Omafilcon A ll 2
Number analyzed (Participants) | 49 | 48 | 49
units on a scale
  Conjunctival Hyperemia | 0.76 (0.26) | 0.79 (0.31) | 0.78 (0.28)
  Limbal Hyperaemia | 0.63 (0.24) | 0.66 (0.30) | 0.65 (0.28)
  Corneal Vascularization | 0.05 (0.11) | 0.05 (0.10) | 0.06 (0.09)
  Microcysts | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00)
  Oedema | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00)
  Corneal Staining | 0.33 (0.42) | 0.42 (0.43) | 0.26 (0.36)
  Conjunctival Staining | 1.37 (0.65) | 0.41 (0.43) | 0.23 (0.20)
  Paipliiary Conjunctivitis | 0.95 (0.28) | 0.88 (0.35) | 0.93 (0.34)

2. Secondary Outcome: Lens Fit - Horizontal Centration
Description: Horizontal centration will be assessed for the following regions: extremely nasal, slightly nasal, optimum, slightly temporal, extremely temporal.
Time Frame: 1 week
Population: Protocol deviations and discontinuations account for difference in analysis population
Measure: Count of Participants; unit: Participants
Arm/Group | Somofilcon A | Nelfilcon A II 2 | Omafilcon A ll 2
Number analyzed (Participants) | 49 | 48 | 49
Participants
  Extremely Nasal | 0 | 0 | 0
  Slightly Nasal | 1 | 3 | 1
  Optimum | 28 | 28 | 26
  Slightly Temporal | 20 | 17 | 22
  Extremely Temporal | 0 | 0 | 0

3. Secondary Outcome: Lens Fit - Vertical Centration
Description: Vertical centration will be assessed for the following regions: extremely nasal, slightly nasal, optimum, slightly temporal, extremely nasal.
Time Frame: 1 week
Population: Protocol deviations and discontinuations account for difference in analysis population
Measure: Count of Participants; unit: Participants
Arm/Group | Somofilcon A | Nelfilcon A II 2 | Omafilcon A ll 2
Number analyzed (Participants) | 49 | 48 | 49
Participants
  Extremely Nasal | 0 | 0 | 0
  Slightly Nasal | 11 | 20 | 22
  Optimum | 21 | 22 | 22
  Slightly Temporal | 17 | 6 | 5
  Extremely Temporal | 0 | 0 | 0

4. Secondary Outcome: Lens Fit - Corneal Coverage
Description: Corneal coverage will be assessed for the following regions: extremely nasal, slightly nasal, optimum, slightly temporal, extremely nasal.
Time Frame: 1 week
Population: Protocol deviations and discontinuations account for difference in analysis population
Measure: Count of Participants; unit: Participants
Arm/Group | Somofilcon A | Nelfilcon A II 2 | Omafilcon A ll 2
Number analyzed (Participants) | 49 | 48 | 49
Participants
  Extremely Nasal | 0 | 0 | 0
  Slightly Nasal | 3 | 7 | 4
  Optimum | 46 | 39 | 41
  Slightly Temporal | 0 | 2 | 4
  Extremely Temporal | 0 | 0 | 0

5. Secondary Outcome: Lens Fit - Movement
Description: Lens movement assessed using the following evaluations: extremely inadequate, slightly inadequate, optimum, slightly excessive, extremely excessive.
Time Frame: 1 week
Population: Protocol deviations and discontinuations account for difference in analysis population
Measure: Count of Participants; unit: Participants
Arm/Group | Somofilcon A | Nelfilcon A II 2 | Omafilcon A ll 2
Number analyzed (Participants) | 49 | 48 | 49
Participants
  Extremely inadequate | 0 | 0 | 0
  Slightly inadequate | 3 | 19 | 12
  Optimum | 38 | 27 | 27
  Slightly excessive | 8 | 2 | 9
  Extremely excessive | 0 | 0 | 1

6. Secondary Outcome: Lens Surface - Deposition
Description: Lens surface will be assessed using Grades 0-4, 0=normal, 1=trace, 2=mild, 3=moderate, 4=severe
Time Frame: 1 week
Population: Protocol deviations and discontinuations account for difference in analysis population
Measure: Count of Participants; unit: Participants
Arm/Group | Somofilcon A | Nelfilcon A II 2 | Omafilcon A ll 2
Number analyzed (Participants) | 49 | 48 | 49
Participants
  Grade 0 | 46 | 47 | 48
  Grade 1 | 3 | 1 | 1
  Grade 2 | 0 | 0 | 0
  Grade 3 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0

7. Secondary Outcome: Lens Surface - Wettability
Description: Lens wettability will be assessed using Grades 0-4, 0=normal, 1=trace, 2=mild, 3=moderate, 4=severe
Time Frame: 1 week
Population: Protocol deviations and discontinuations account for difference in analysis population
Measure: Count of Participants; unit: Participants
Arm/Group | Somofilcon A | Nelfilcon A II 2 | Omafilcon A ll 2
Number analyzed (Participants) | 49 | 48 | 49
Participants
  Grade 0 | 37 | 44 | 43
  Grade 1 | 9 | 3 | 3
  Grade 2 | 3 | 1 | 3
  Grade 3 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0

8. Secondary Outcome: Visual Acuity
Description: Visual acuity will be assessed by LogMAR.
Time Frame: 1 week
Population: Protocol deviations and discontinuations account for difference in analysis population
Measure: Mean (Standard Deviation); unit: LogMAR
Arm/Group | Somofilcon A | Nelfilcon A II 2 | Omafilcon A ll 2
Number analyzed (Participants) | 49 | 48 | 49
LogMAR
  High Contrast | -0.11 (0.08) | -0.13 (0.08) | -0.11 (0.07)
  Low Contrast | 0.18 (0.10) | 0.17 (0.11) | 0.18 (0.10)

ADVERSE EVENTS:
Time Frame: Subjects were randomized to wear each pair of lenses (Somofilcon A, Nelfilcon A II 2, Omafilcon A II 2 at a random sequence) for One- Week in a random sequence, assessed overall for up to 4 weeks.
Groups:
- Somofilcon A: Subjects are randomized to wear Somofilcon A for one week at random sequence
- Nelfilcon A II 2: Subjects are randomized to wear Nelfilcon A II 2 for one week at random sequence
- Omafilcon A II 2: Subjects are randomized to wear Omafilcon A II 2 for one week at random sequence
Arm/Group | Somofilcon A | Nelfilcon A II 2 | Omafilcon A II 2
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/48 | 0/49
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/48 | 0/49
Other Adverse Events (participants affected / at risk) | 4/49 | 3/48 | 4/49
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Somofilcon A (N=49) | Nelfilcon A II 2 (N=48) | Omafilcon A II 2 (N=49)
Common cold (Infections and infestations) | 4 (4) | 3 (3) | 4 (4) — Non-ocular adverse events reported during the study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes